CLINICAL TRIAL: NCT02144584
Title: Pilot Study of Memantine for Enhanced Stroke Recovery
Brief Title: Memantine for Enhanced Stroke Recovery
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Jennifer Majersik, M.D, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00068751
Record Dates: First submitted 2014-01-27; First posted 2014-05-22 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Ischemic Stroke; Upper Extremity Weakness
Keywords: ischemic stroke; memantine; upper extremity weakness; motor recovery
MeSH Terms: conditions — Ischemic Stroke; Paresis | interventions — Memantine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo plus standard of care (Placebo Comparator): Participants will start taking either memantine or placebo within 24 hours after baseline testing and randomization is completed, but no later than day 8 post-symptom onset. Participants will titrate up on the dose of placebo until taking twice daily. Participants will continue for 90 days with placebo. Continue with standard of care for other treatment of stroke.
  Interventions: Drug: Placebo (for memantine)
- Memantine plus standard of care (Active Comparator): Participants will start taking either memantine or placebo within 24 hours after baseline testing and randomization is completed, but no later than day 8 post-symptom onset. Participants will use a titration schedule starting at 7mg daily for 1 week, increasing by 7mg (1 capsule) per week until at a goal dose of 28mg daily (goal dose) as recommend by the manufacturer. Participants will continue memantine for 90 days. Continue with standard care for stroke.
  Interventions: Drug: Memantine XR

INTERVENTIONS:
Drug: Memantine XR — The active drug will be encapsulated by the University of Utah Research Pharmacy to maintain blinding.
  Other Names: Namenda XR
  Arms: Memantine plus standard of care
Drug: Placebo (for memantine) — Placebo to be capsuled to look identical to active drug (memantine)
  Other Names: sugar capsule
  Arms: Placebo plus standard of care

SUMMARY:
This will be a randomized double blind placebo-controlled pilot study using a repeated measures design in which participants with acute ischemic stroke and upper extremity weakness are randomized to either drug or placebo

DETAILED DESCRIPTION:
This will be a randomized double blind placebo-controlled pilot study using a repeated measures design in which participants with acute ischemic stroke and upper extremity weakness are randomized to either drug or placebo, complete therapy, and complete outcomes assessments at baseline, 4, and 12 weeks post-stroke. Target enrollment will be 10 patients per group and adaptive randomization will be used to assist with equal representation of pre-stroke selective serotonin reuptake inhibitor (SSRI) use and motor severity (Fugl-Meyer score) in each arm. The primary purpose of this pilot study is to measure adverse events, drop-out rates, feasibility of trial conductance, and establishment of effect sizes in each group in order to power a larger efficacy trial at the University of Utah. An intention to treat model will be used during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years old
2. Randomization between 3 days-8 weeks days of stroke symptom onset
3. Arm weakness severe enough to warrant inpatient or outpatient occupational therapies
4. Able to voluntarily move affected UE
5. Living independently prior to their stroke
6. Image-confirmed ischemic stroke (MRI or CT)
7. Supratentorial location of stroke
8. Fugl-Meyer Upper Extremity Score of 50 or less and/or Fugl Meyer Lower Extremity Score of 28 or less
9. Ability to swallow pills

Exclusion Criteria:

1. subarachnoid hemorrhage, subdural hemorrhage or other cause of symptoms other than ischemic or hemorrhagic stroke
2. Infratentorial location of stroke (brainstem or cerebellum)
3. NIH Stroke Scale >20 at the time of randomization
4. History of dementia that will interfere with rehabilitation
5. Pre or post-stroke use of memantine or amantadine
6. Contraindications to taking memantine XR in pill form
7. History of prior clinical stroke with residual symptoms on the same side as the current symptoms that would interfere with outcomes of this study
8. Documented severe renal impairment (CrCl < 30 ml/min) Blood tests will be performed prior to study procedures that will ensure patients do not have renal impairment if not done as part of clinical care.
9. Moribund or not expected to live 6 months
10. Severe cognitive deficits or pre-morbid function causing inaccurate neurologic assessment or inability to complete the initial assessment
11. Comorbid neurologic disease that would interfere with the results including but not limited to Multiple Sclerosis, neurodegenerative diseases, spinal cord disease, and central nervous system cancer.
12. Documented severe hepatic impairment (Child-Pugh score > 6) or severe hepatic disease (hepatitis)
13. Patients who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment | 30 days
  Fugl-Meyer Assessment UE and LE scales (FMUE and FMLE). Our primary outcome measures will be the scores on the FMUE and FMLE as they have been shown to have good reliability and validity.
  These scales measure motor impairment by asking the participant to perform various arm, hand, and leg motions. Items are scored on a 3-point scale with 0 representing no movement, 1 representing the inability to complete the entire item and 2 representing ability to complete the item as asked. Scores range from 0-66 on the FMUE and 0-34 on the FMLE with higher scores indicating better motor control. In addition, the proprioception subscale of the FM will be used to assess status of proprioception in the UE and LE. The hip, knee, ankle, big toe, shoulder, elbow, wrist, and the thumb are moved passively and the participant is asked to indicate in which direction the joint was moved.
Fugl-Meyer Assessment | 90 days
  Fugl-Meyer Assessment UE and LE scales (FMUE and FMLE). Our primary outcome measures will be the scores on the FMUE and FMLE as they have been shown to have good reliability and validity.
  These scales measure motor impairment by asking the participant to perform various arm, hand, and leg motions. Items are scored on a 3-point scale with 0 representing no movement, 1 representing the inability to complete the entire item and 2 representing ability to complete the item as asked. Scores range from 0-66 on the FMUE and 0-34 on the FMLE with higher scores indicating better motor control. In addition, the proprioception subscale of the FM will be used to assess status of proprioception in the UE and LE. The hip, knee, ankle, big toe, shoulder, elbow, wrist, and the thumb are moved passively and the participant is asked to indicate in which direction the joint was moved.
Adverse events | up to 30 days
  Participants will be contacted by the stroke research nurse after weeks 1, 2, 3, and 8 of after randomization by telephone call or inpatient visit (if in the hospital or acute inpatient rehabilitation). Participants will be asked about potential adverse events during each phone call and each clinic visit. All adverse events, serious and minor, will be recorded on an adverse event table. The study investigators will review study records after every 5 participants are enrolled to monitor for patterns of adverse events to evaluate the safety of continuing the study.
Adverse Events | 30-90 days
  Participants will be contacted by the stroke research nurse after weeks 1, 2, 3, and 8 of after randomization by telephone call or inpatient visit (if in the hospital or acute inpatient rehabilitation). Participants will be asked about potential adverse events during each phone call and each clinic visit. All adverse events, serious and minor, will be recorded on an adverse event table. The study investigators will review study records after every 5 participants are enrolled to monitor for patterns of adverse events to evaluate the safety of continuing the study.

SECONDARY OUTCOMES:
Motor Activity Log (MAL) | 30 days
  The validity of the MAL has been well established against upper extremity accelerometry.
  The Motor Activity Log is a self-report measure of how frequently the participant uses his or her paretic hand in 30 common daily activities, such as opening a drawer and shaving or putting on make-up. Participants rate how often they use the paretic UE in these tasks on a 6 point scale from 0 representing no use to 5 representing as much use as before the stroke. The quality of movement scale on the Motor Activity Log asks the participant to rate how well he or she perceives the task is performed with the paretic UE. The ratings are also made on a 6 point scale with 0 representing no use to 5 representing as well as before the stroke. This assessment will only be completed at post-intervention and follow-up as it is invalid assessment in the in-patient setting where participants have few opportunities to engage in the tested items.
Motor Activity Log (MAL) | 90 days
  The validity of the MAL has been well established against upper extremity accelerometry.
  The Motor Activity Log is a self-report measure of how frequently the participant uses his or her paretic hand in 30 common daily activities, such as opening a drawer and shaving or putting on make-up. Participants rate how often they use the paretic UE in these tasks on a 6 point scale from 0 representing no use to 5 representing as much use as before the stroke. The quality of movement scale on the Motor Activity Log asks the participant to rate how well he or she perceives the task is performed with the paretic UE. The ratings are also made on a 6 point scale with 0 representing no use to 5 representing as well as before the stroke. This assessment will only be completed at post-intervention and follow-up as it is invalid assessment in the in-patient setting where participants have few opportunities to engage in the tested items.
Ten Meter Walk Test | 30 days
  The 10 meter walk is a measure of typical gait speed.
  The participant is asked to walk at his/her usual pace for 10 meters along a hallway. Two trials are completed with the best time in seconds to walk the distance recorded. The test is reliable. We will videotape the walk and later use the Riverside Scale for rating quality of locomotion.
Ten Meter Walk Test | 90 days
  The 10 meter walk is a measure of typical gait speed.
  The participant is asked to walk at his/her usual pace for 10 meters along a hallway. Two trials are completed with the best time in seconds to walk the distance recorded. The test is reliable. We will videotape the walk and later use the Riverside Scale for rating quality of locomotion.
Stroke Impact Scale (SIS) | 30 days
  The SIS is a self-report measure of functioning after stroke at the body function, activity, and participation levels.
  Participants rate on a 5 point scale how frequently statements apply to them across 8 domains (strength, communication, emotion, hand use, activities of daily living, mobility, thinking, and social participation). Scores for each domain are tallied and converted to a 100-point scale. Scores across domains are also tallied and converted to a 100-point scale. The SIS has been shown to be reliable and valid. This assessment will only be completed at post-intervention and follow-up as many of the items concern activities that are only encountered in the community. Participants who are new inpatients will not have had the opportunity to engage in these activities.
Stroke Impact Scale (SIS) | 90 days
  The SIS is a self-report measure of functioning after stroke at the body function, activity, and participation levels.
  Participants rate on a 5 point scale how frequently statements apply to them across 8 domains (strength, communication, emotion, hand use, activities of daily living, mobility, thinking, and social participation). Scores for each domain are tallied and converted to a 100-point scale. Scores across domains are also tallied and converted to a 100-point scale. The SIS has been shown to be reliable and valid. This assessment will only be completed at post-intervention and follow-up as many of the items concern activities that are only encountered in the community. Participants who are new inpatients will not have had the opportunity to engage in these activities.
Cancellation Tests | 30 Days
  These tests measure the presence of unilateral neglect.
  The letter cancellation task includes 40 target letters (E, R) among 130 non-target letters on an A4-sized landscape sheet (maximum score 40, cutoff point 32). The letters are arranged in five rows, each containing 34 items. The star cancellation task consists of 56 targets (small stars) and 75 non-targets (big stars, words, and letters) randomly spaced on an A4-sized landscape sheet. In these three cancellation tasks, participants are instructed to search and mark all the targets on the stimulus sheet. The total number of targets crossed out on the left and the right of each form will be tallied and the percentage.
Cancellations Tests | 90 Days
  These tests measure the presence of unilateral neglect.
  The letter cancellation task includes 40 target letters (E, R) among 130 non-target letters on an A4-sized landscape sheet (maximum score 40, cutoff point 32). The letters are arranged in five rows, each containing 34 items. The star cancellation task consists of 56 targets (small stars) and 75 non-targets (big stars, words, and letters) randomly spaced on an A4-sized landscape sheet. In these three cancellation tasks, participants are instructed to search and mark all the targets on the stimulus sheet. The total number of targets crossed out on the left and the right of each form will be tallied and the percentage.
Grip Strength Test | 30 Days
  Grip strength will be tested using the American Hand Therapy Association recommended protocol.
  Briefly, the participant will be seated in a straight backed chair with the paretic shoulder in neutral, elbow flexed, forearm half-way between supination and pronation. He or she grasps the Jamar-type dynamometer by the handle and squeezes it as hard as possible for 5 seconds. The tester gives the command "Ok, squeeze as hard as you can….harder…..harder…..relax". The test is repeated 2 more times with a 30 second rest in between squeezes. Grip strength will be measured as the average of the 3 trials to the nearest kilogram.
Grip Strength Test | 90 Days
  Grip strength will be tested using the American Hand Therapy Association recommended protocol.
  Briefly, the participant will be seated in a straight backed chair with the paretic shoulder in neutral, elbow flexed, forearm half-way between supination and pronation. He or she grasps the Jamar-type dynamometer by the handle and squeezes it as hard as possible for 5 seconds. The tester gives the command "Ok, squeeze as hard as you can….harder…..harder…..relax". The test is repeated 2 more times with a 30 second rest in between squeezes. Grip strength will be measured as the average of the 3 trials to the nearest kilogram.
Montreal Cognitive Assessment (MoCA©) | 30 Days
  The MoCA© is recommended by NIH and Canadian Stroke Consortium for Cognitive Assessment after Stroke. It is reliable and valid for the stroke population.
Montreal Cognitive Assessment (MoCA©) | 90 Days
  The MoCA© is recommended by NIH and Canadian Stroke Consortium for Cognitive Assessment after Stroke. It is reliable and valid for the stroke population.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Bennett, D.O., Principal Investigator — University of Utah; Jennifer Majersik, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Magid D, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER, Moy CS, Mussolino ME, Nichol G, Paynter NP, Schreiner PJ, Sorlie PD, Stein J, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Executive summary: heart disease and stroke statistics--2013 update: a report from the American Heart Association. Circulation. 2013 Jan 1;127(1):143-52. doi: 10.1161/CIR.0b013e318282ab8f. No abstract available. PMID 23283859
- [Background] Rathore SS, Hinn AR, Cooper LS, Tyroler HA, Rosamond WD. Characterization of incident stroke signs and symptoms: findings from the atherosclerosis risk in communities study. Stroke. 2002 Nov;33(11):2718-21. doi: 10.1161/01.str.0000035286.87503.31. PMID 12411667
- [Background] Kalra L, Eade J. Role of stroke rehabilitation units in managing severe disability after stroke. Stroke. 1995 Nov;26(11):2031-4. doi: 10.1161/01.str.26.11.2031. PMID 7482644
- [Background] Chollet F, Tardy J, Albucher JF, Thalamas C, Berard E, Lamy C, Bejot Y, Deltour S, Jaillard A, Niclot P, Guillon B, Moulin T, Marque P, Pariente J, Arnaud C, Loubinoux I. Fluoxetine for motor recovery after acute ischaemic stroke (FLAME): a randomised placebo-controlled trial. Lancet Neurol. 2011 Feb;10(2):123-30. doi: 10.1016/S1474-4422(10)70314-8. Epub 2011 Jan 7. PMID 21216670
- [Background] Ziemann U, Ilic TV, Pauli C, Meintzschel F, Ruge D. Learning modifies subsequent induction of long-term potentiation-like and long-term depression-like plasticity in human motor cortex. J Neurosci. 2004 Feb 18;24(7):1666-72. doi: 10.1523/JNEUROSCI.5016-03.2004. PMID 14973238
- [Background] Lipton SA. Failures and successes of NMDA receptor antagonists: molecular basis for the use of open-channel blockers like memantine in the treatment of acute and chronic neurologic insults. NeuroRx. 2004 Jan;1(1):101-10. doi: 10.1602/neurorx.1.1.101. PMID 15717010
- [Background] Chen HS, Lipton SA. Mechanism of memantine block of NMDA-activated channels in rat retinal ganglion cells: uncompetitive antagonism. J Physiol. 1997 Feb 15;499 ( Pt 1)(Pt 1):27-46. doi: 10.1113/jphysiol.1997.sp021909. PMID 9061638
- [Background] Chen HS, Pellegrini JW, Aggarwal SK, Lei SZ, Warach S, Jensen FE, Lipton SA. Open-channel block of N-methyl-D-aspartate (NMDA) responses by memantine: therapeutic advantage against NMDA receptor-mediated neurotoxicity. J Neurosci. 1992 Nov;12(11):4427-36. doi: 10.1523/JNEUROSCI.12-11-04427.1992. PMID 1432103
- [Background] Chen HS, Wang YF, Rayudu PV, Edgecomb P, Neill JC, Segal MM, Lipton SA, Jensen FE. Neuroprotective concentrations of the N-methyl-D-aspartate open-channel blocker memantine are effective without cytoplasmic vacuolation following post-ischemic administration and do not block maze learning or long-term potentiation. Neuroscience. 1998 Oct;86(4):1121-32. doi: 10.1016/s0306-4522(98)00163-8. PMID 9697119
- [Background] Parsons CG, Danysz W, Quack G. Memantine is a clinically well tolerated N-methyl-D-aspartate (NMDA) receptor antagonist--a review of preclinical data. Neuropharmacology. 1999 Jun;38(6):735-67. doi: 10.1016/s0028-3908(99)00019-2. PMID 10465680
- [Background] Kilic U, Yilmaz B, Reiter RJ, Yuksel A, Kilic E. Effects of memantine and melatonin on signal transduction pathways vascular leakage and brain injury after focal cerebral ischemia in mice. Neuroscience. 2013 May 1;237:268-76. doi: 10.1016/j.neuroscience.2013.01.059. Epub 2013 Feb 8. PMID 23396088
- [Background] LUCAS DR, NEWHOUSE JP. The toxic effect of sodium L-glutamate on the inner layers of the retina. AMA Arch Ophthalmol. 1957 Aug;58(2):193-201. doi: 10.1001/archopht.1957.00940010205006. No abstract available. PMID 13443577
- [Background] Leveille F, El Gaamouch F, Gouix E, Lecocq M, Lobner D, Nicole O, Buisson A. Neuronal viability is controlled by a functional relation between synaptic and extrasynaptic NMDA receptors. FASEB J. 2008 Dec;22(12):4258-71. doi: 10.1096/fj.08-107268. Epub 2008 Aug 18. PMID 18711223
- [Background] Wenk GL, Zajaczkowski W, Danysz W. Neuroprotection of acetylcholinergic basal forebrain neurons by memantine and neurokinin B. Behav Brain Res. 1997 Feb;83(1-2):129-33. doi: 10.1016/s0166-4328(97)86056-1. PMID 9062671
- [Background] Palmer GC. Neuroprotection by NMDA receptor antagonists in a variety of neuropathologies. Curr Drug Targets. 2001 Sep;2(3):241-71. doi: 10.2174/1389450013348335. PMID 11554551
- [Background] Babu CS, Ramanathan M. Pre-ischemic treatment with memantine reversed the neurochemical and behavioural parameters but not energy metabolites in middle cerebral artery occluded rats. Pharmacol Biochem Behav. 2009 May;92(3):424-32. doi: 10.1016/j.pbb.2009.01.010. Epub 2009 Jan 23. PMID 19463256
- [Background] Cho GS, Lee JC, Ju C, Kim C, Kim WK. N-Methyl-D-aspartate receptor antagonists memantine and MK-801 attenuate the cerebral infarct accelerated by intracorpus callosum injection of lipopolysaccharides. Neurosci Lett. 2013 Mar 22;538:9-14. doi: 10.1016/j.neulet.2013.01.031. Epub 2013 Jan 30. PMID 23376060
- [Background] Culmsee C, Junker V, Kremers W, Thal S, Plesnila N, Krieglstein J. Combination therapy in ischemic stroke: synergistic neuroprotective effects of memantine and clenbuterol. Stroke. 2004 May;35(5):1197-202. doi: 10.1161/01.STR.0000125855.17686.6d. Epub 2004 Apr 1. PMID 15060319
- [Background] Lapchak PA. Memantine, an uncompetitive low affinity NMDA open-channel antagonist improves clinical rating scores in a multiple infarct embolic stroke model in rabbits. Brain Res. 2006 May 9;1088(1):141-7. doi: 10.1016/j.brainres.2006.02.093. Epub 2006 Apr 13. PMID 16626666
- [Background] Montagne A, Hebert M, Jullienne A, Lesept F, Le Behot A, Louessard M, Gauberti M, Orset C, Ali C, Agin V, Maubert E, Vivien D. Memantine improves safety of thrombolysis for stroke. Stroke. 2012 Oct;43(10):2774-81. doi: 10.1161/STROKEAHA.112.669374. Epub 2012 Aug 9. PMID 22879098
- [Background] Tariot PN, Farlow MR, Grossberg GT, Graham SM, McDonald S, Gergel I; Memantine Study Group. Memantine treatment in patients with moderate to severe Alzheimer disease already receiving donepezil: a randomized controlled trial. JAMA. 2004 Jan 21;291(3):317-24. doi: 10.1001/jama.291.3.317. PMID 14734594
- [Background] Emre M, Tsolaki M, Bonuccelli U, Destee A, Tolosa E, Kutzelnigg A, Ceballos-Baumann A, Zdravkovic S, Bladstrom A, Jones R; 11018 Study Investigators. Memantine for patients with Parkinson's disease dementia or dementia with Lewy bodies: a randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2010 Oct;9(10):969-77. doi: 10.1016/S1474-4422(10)70194-0. Epub 2010 Aug 20. PMID 20729148
- [Background] Iwamoto K, Ikeda K, Mizumura S, Tachiki K, Yanagihashi M, Iwasaki Y. Combined treatment of methylprednisolone pulse and memantine hydrochloride prompts recovery from neurological dysfunction and cerebral hypoperfusion in carbon monoxide poisoning: a case report. J Stroke Cerebrovasc Dis. 2014 Mar;23(3):592-5. doi: 10.1016/j.jstrokecerebrovasdis.2013.05.014. Epub 2013 Jun 19. PMID 23791468
- [Background] Berthier ML, Green C, Lara JP, Higueras C, Barbancho MA, Davila G, Pulvermuller F. Memantine and constraint-induced aphasia therapy in chronic poststroke aphasia. Ann Neurol. 2009 May;65(5):577-85. doi: 10.1002/ana.21597. PMID 19475666
- [Background] Fugl-Meyer AR, Jaasko L, Leyman I, Olsson S, Steglind S. The post-stroke hemiplegic patient. 1. a method for evaluation of physical performance. Scand J Rehabil Med. 1975;7(1):13-31. PMID 1135616
- [Background] Duncan PW, Propst M, Nelson SG. Reliability of the Fugl-Meyer assessment of sensorimotor recovery following cerebrovascular accident. Phys Ther. 1983 Oct;63(10):1606-10. doi: 10.1093/ptj/63.10.1606. PMID 6622535
- [Background] Taub E, Miller NE, Novack TA, Cook EW 3rd, Fleming WC, Nepomuceno CS, Connell JS, Crago JE. Technique to improve chronic motor deficit after stroke. Arch Phys Med Rehabil. 1993 Apr;74(4):347-54. PMID 8466415
- [Background] van der Lee JH, Beckerman H, Knol DL, de Vet HC, Bouter LM. Clinimetric properties of the motor activity log for the assessment of arm use in hemiparetic patients. Stroke. 2004 Jun;35(6):1410-4. doi: 10.1161/01.STR.0000126900.24964.7e. Epub 2004 Apr 15. PMID 15087552
- [Background] Uswatte G, Taub E, Morris D, Light K, Thompson PA. The Motor Activity Log-28: assessing daily use of the hemiparetic arm after stroke. Neurology. 2006 Oct 10;67(7):1189-94. doi: 10.1212/01.wnl.0000238164.90657.c2. PMID 17030751
- [Background] Collen FM, Wade DT, Bradshaw CM. Mobility after stroke: reliability of measures of impairment and disability. Int Disabil Stud. 1990 Jan-Mar;12(1):6-9. doi: 10.3109/03790799009166594. PMID 2211468
- [Background] Duncan PW, Wallace D, Lai SM, Johnson D, Embretson S, Laster LJ. The stroke impact scale version 2.0. Evaluation of reliability, validity, and sensitivity to change. Stroke. 1999 Oct;30(10):2131-40. doi: 10.1161/01.str.30.10.2131. PMID 10512918
- [Background] Kidd D, Stewart G, Baldry J, Johnson J, Rossiter D, Petruckevitch A, Thompson AJ. The Functional Independence Measure: a comparative validity and reliability study. Disabil Rehabil. 1995 Jan;17(1):10-4. doi: 10.3109/09638289509166622. PMID 7858276